CLINICAL TRIAL: NCT07154485
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, Investigator-initiated Phase 2a Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics (PK/PD), and Exploratory Efficacy of Multiple Doses of NS101 in Patients With Semantic Variant Primary Progressive Aphasia (svPPA), a Subtype of Frontotemporal Dementia (FTD)
Brief Title: Investigator Initiated Study for the Safety and Efficacy in Frontotemporal Dementia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hee-Jin Kim (Other)
Collaborators: Asan Medical Center (Other); Gangnam Severance Hospital (Other); Konkuk University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Hee-Jin Kim, Professor, Department of Neurology, College of Medicine, Hanyang university, Hanyang University Seoul Hospital
Organization: Hanyang University Seoul Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS101_I2a_FTD
Record Dates: First submitted 2025-08-12; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Dementia Frontotemporal
Keywords: Frontotemporal Dementia; semantic variant; FTD; sv FTD; PPA; sv PPA
MeSH Terms: conditions — Pick Disease of the Brain; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NS101 Treatment Group (Active Comparator): Participants will receive a two loading dose of NS101 15 mg/kg IV infusion, followed by biweekly dosing for 6 months during the double-blind phase. Those who complete the double-blind phase will be eligible to enter a 3-month open-label extension to receive active treatment.
  Interventions: Drug: NS101 IV infusion
- NS101 Placebo Group (Placebo Comparator): Participants will receive a two loading dose of NS101 15 mg/kg IV infusion, followed by biweekly dosing for 6 months during the double-blind phase. Those who complete the double-blind phase will be eligible to enter a 3-month open-label extension to receive active treatment.
  Interventions: Drug: Placebo IV Infusion

INTERVENTIONS:
Drug: NS101 IV infusion — NS101 is anti FAM19A5 antibody expected to play as a synapse organizer and reversing synapse dysfunction in various neurological diseases
  Arms: NS101 Treatment Group
Drug: Placebo IV Infusion — Placebo (i.e. fake drug without active pharmaceutical ingredient) of NS101
  Arms: NS101 Placebo Group

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics (PK/PD), immunogenicity, and efficacy of multiple intravenous administrations of the investigational drug NS101, compared to placebo, in patients with semantic variant primary progressive aphasia (svPPA), a subtype of frontotemporal dementia (FTD)

ELIGIBILITY:
Key Inclusion Criteria:

* Participants diagnosed at screening with mild to moderate frontotemporal dementia, semantic variant (svFTD), defined by a CDR® Plus NACC FTLD Sum of Boxes (SOB) score between 4.5 and 15.5.
* Participants confirmed to be amyloid-negative based on Amyloid PET scan or CSF results within the past 36 months.

Key Exclusion Criteria:

* Participants with other degenerative brain diseases as determined by the investigator
* Participants with other neurological disorders and uncontrolled acute disease

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (Safety and Tolerability) | Every Visit for 12month(48weeks)
  To evaluate the safety and tolerability of repeated administration of NS101 compared to placebo in patients with semantic variant primary progressive aphasia (svPPA), a subtype of frontotemporal dementia (FTD).
  <primary efficacy endpoint> The incidence, causality, and severity of adverse events (AEs), serious adverse events (SAEs), adverse drug reactions (ADRs), and serious adverse drug reactions (SADRs) by group.

SECONDARY OUTCOMES:
Plasma FAM19A5 Concentration | Every Visit for 12month(48weeks)
  To assess the pharmacodynamic (PD) effect of NS101 compared to placebo in patients with svPPA
Minimum Plasma Concentration of NS101 (Cmin, Ctrough) | Every Visit for 12month(48weeks)
  To evaluate the pharmacokinetics (PK) of repeated administration of NS101 compared to placebo in patients with svPPA
Anti-Drug Antibodies (ADA) | Every Visit for 12month(48weeks
  To evaluate immunogenicity following repeated administration of NS101 compared to placebo
Neutralizing Antibodies (NAbs) | Every Visit for 12month(48weeks)
  To evaluate the presence of neutralizing antibodies following repeated administration of NS101 compared to placebo

OTHER OUTCOMES:
Change From Baseline in Neuropsychological Test Scores (FAB) | Changes from baseline at each assessment time point - Screening, Week 24, Week 36, Week48
  Neuropsychological assessment
  - Score on Frontal Assessment Battery (FAB)
Change from Baseline in Biomarkers | Changes from baseline at each assessment time point • Screening, Week 24, Week 36, Week48
  Biomarkers
  * Concentration of Neurofilament Light Chain (NfL) [pg/mL]
  * Concentration of Glial Fibrillary Acidic Protein (GFAP) [pg/mL]
Change from Baseline in Brain MRI | Changes from baseline at each assessment time point • Screening, Week 24, Week 36, Week48
  Neuroimaging
  - Brain MRI Measures With Functional MRI (fMRI)
Change From Baseline in Neuropsychological Test Scores (BNT/WAB) | Changes from baseline at each assessment time point - Screening, Week 24, Week 36, Week48
  Neuropsychological assessment
  - Score on Boston Naming Test (BNT) or Western Aphasia Battery (WAB)
Change From Baseline in Neuropsychological Test Scores (ADCS-ADL) | Changes from baseline at each assessment time point - Screening, Week 24, Week 36, Week48
  Neuropsychological assessment
  - Score on Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
Change From Baseline in Neuropsychological Test Scores (FBI) | Changes from baseline at each assessment time point - Screening, Week 24, Week 36, Week48
  Neuropsychological assessment
  - Score on Frontal Behavioral Inventory (FBI)
Change From Baseline in Neuropsychological Test Scores (C-SSRS) | Changes from baseline at each assessment time point - Screening, Week 24, Week 36, Week48
  Neuropsychological assessment
  - Score on Columbia-Suicide Severity Rating Scale (C-SSRS)

IPD SHARING:
Plan to Share IPD: No